CLINICAL TRIAL: NCT02633410
Title: Prospective Randomized Clinical Study Comparing Anteromedial Portal Versus Transtibial Technique for Femoral Tunnel Positioning in Anterior Cruciate Ligament Reconstruction With Hamstring Autograft
Brief Title: Transtibial Versus Anteromedial Femoral Tunnel Technique in ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACL-FEM 01
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transtibial (Active Comparator): Transtibial technique used to create femoral tunnel
  Interventions: Procedure: Femoral tunnel creation
- Anteromedial (Active Comparator): Anteromedial technique used to create femoral tunnel
  Interventions: Procedure: Femoral tunnel creation

INTERVENTIONS:
Procedure: Femoral tunnel creation — Arthroscopic surgery approach used to create tunnel in femur into which graft is positioned

SUMMARY:
The anteromedial (AM) portal technique was introduced to position the femoral tunnel in anterior cruciate ligament (ACL) reconstruction to more closely replicate the original footprint compared to the transtibial (TT) approach.1-5 Few randomized trials have evaluated differences in these techniques with respect to clinical outcomes. The purpose of this study was to determine if there are any differences in clinical outcome between the AM and TT approaches.

DETAILED DESCRIPTION:
The anteromedial (AM) portal technique was introduced to position the femoral tunnel in anterior cruciate ligament (ACL) reconstruction to more closely replicate the original footprint compared to the transtibial (TT) approach.1-5 Few randomized trials have evaluated differences in these techniques with respect to clinical outcomes. The purpose of this study was to determine if there are any differences in clinical outcome between the AM and TT approaches.

ELIGIBILITY:
Inclusion Criteria:

* sustained a complete ACL tear and had no other ligament injuries requiring surgical intervention

Exclusion Criteria:

* concomitant collateral ligament tears
* significant chondromalacia (based on diagnostic imaging)
* previous lower limb surgery
* significant injury to either lower limb requiring surgery
* history of arthritis
* were unable to comply with rehabilitation protocols or study follow-ups
* were pregnant females or had other medical conditions which precluded participation.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2007-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Anterior cruciate ligament quality of life | 24-months postoperative

SECONDARY OUTCOMES:
KT-1000 | 24-months post-operative
Knee range of motion | 24-months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Peter MacDonald, MD FRCSC, Principal Investigator — Pan Am CLinic/University of Manitoba